CLINICAL TRIAL: NCT03037840
Title: Detecting Tumor Specific Amplitude-modulated Frequencies of Cancer Patients In Vivo
Brief Title: Detecting Tumor Specific Amplitude-modulated Frequencies of Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southern Medical University, China (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Guangdong 999 Brain Hospital (Other); The 157th Hospital of PLA,China (Unknown)
Responsible Party: Principal Investigator, Sherman Xuegang Xin, Professor, Southern Medical University, China
Other Study IDs: SXXin-AM-RF-EMF-in vivo
Record Dates: First submitted 2016-07-06; First posted 2017-01-31 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Neoplasms
Keywords: RF EMF; In Vivo; tumor specific frequencies
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cancer patients: Low intensity amplitude-modulated RF EMFs
  Interventions: Device: Low intensity amplitude-modulated RF EMFs
- healthy participators: Low intensity amplitude-modulated RF EMFs
  Interventions: Device: Low intensity amplitude-modulated RF EMFs

INTERVENTIONS:
Device: Low intensity amplitude-modulated RF EMFs — Low intensity amplitude-modulated radiofrequency electromagnetic fields,the carrier frequency is 27.12MHz with a power of about 100mW
  Other Names: Low intensity AM RF EMFs

SUMMARY:
Studies have shown that tumor specific amplitude-modulated frequencies of radiofrequency electromagnetic fields that is associated with biofeedback upon exposure to in cancer patients. However, such discovery in other cancer patients are rare. And whether tumor specific frequencies can be found in Asian cancer patients remains unclear. The purpose of this study is to detect the tumor specific frequencies of Asian cancer patients in vivo.

DETAILED DESCRIPTION:
The measurements were safety guaranteed and were conducted in hospital. Before detecting, the patient will be already diagnosed with cancer. The doctor and the operator are responsible for the detecting. When cancer patients are exposure to the RF electromagnetic fields, the radial pulse amplitude, blood pressure, skin electrical resistance and breath will be monitored. Biofeedback parameters will be recorded at different modulation frequencies and analyzed in order to find the variation and tumor specific frequencies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cancer Disease

Exclusion Criteria:

* other patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. The patients who are diagnosed with cancer disease
  2. Healthy participators
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Biofeedback response of cancer patients at the exposure of Low intensity amplitude-modulated radiofrequency electromagnetic fields | within 20 min of exposure

SECONDARY OUTCOMES:
Representation of autonomous response during the exposure of tumor specific frequencies modutated RF eletromagnetic fields | within 20 min of exposure

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sherman Xuegang, professor, Principal Investigator — School of Biomedical Engineering,Southern Medical University; Cai Linbo, master, Study Director — Guangdong 999 Brain Hospital; Zhu Xiaoxia, PhD, Study Director — Nanfang Hospital, Southern Medical University; Liu Xiantang, bachelor, Study Director — The 157th Hospital of PLA

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barbault A, Costa FP, Bottger B, Munden RF, Bomholt F, Kuster N, Pasche B. Amplitude-modulated electromagnetic fields for the treatment of cancer: discovery of tumor-specific frequencies and assessment of a novel therapeutic approach. J Exp Clin Cancer Res. 2009 Apr 14;28(1):51. doi: 10.1186/1756-9966-28-51. PMID 19366446
- [Background] Costa FP, de Oliveira AC, Meirelles R, Machado MC, Zanesco T, Surjan R, Chammas MC, de Souza Rocha M, Morgan D, Cantor A, Zimmerman J, Brezovich I, Kuster N, Barbault A, Pasche B. Treatment of advanced hepatocellular carcinoma with very low levels of amplitude-modulated electromagnetic fields. Br J Cancer. 2011 Aug 23;105(5):640-8. doi: 10.1038/bjc.2011.292. Epub 2011 Aug 9. PMID 21829195
- [Background] Zimmerman JW, Pennison MJ, Brezovich I, Yi N, Yang CT, Ramaker R, Absher D, Myers RM, Kuster N, Costa FP, Barbault A, Pasche B. Cancer cell proliferation is inhibited by specific modulation frequencies. Br J Cancer. 2012 Jan 17;106(2):307-13. doi: 10.1038/bjc.2011.523. Epub 2011 Dec 1. PMID 22134506
- [Background] Zimmerman JW, Jimenez H, Pennison MJ, Brezovich I, Morgan D, Mudry A, Costa FP, Barbault A, Pasche B. Targeted treatment of cancer with radiofrequency electromagnetic fields amplitude-modulated at tumor-specific frequencies. Chin J Cancer. 2013 Nov;32(11):573-81. doi: 10.5732/cjc.013.10177. PMID 24206915